CLINICAL TRIAL: NCT04917900
Title: Single-arm, Multi-center Clinical Study of Pyrotinib Maleate Tablets Combined With Albumin-bound Paclitaxel and Trastuzumab in Neoadjuvant Treatment of Her2-positive Early or Locally Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Shuangyue Liu, Head and Neck Oncology, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-SC-BB-BC-II-010
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: Her2-positve Breast Cancer; Neoadjuvant Therapy; Pyrotinib
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib combined with albumin-bound paclitaxel and trastuzumab (Experimental): Pyrotinib: 400mg, po,qd,with warm water within 30 minutes after breakfast, q3weeks, 6 cycles in total. Albumin-bound paclitaxel: 260mg/m2, iv, Day1, q3weeks, 6 cycles in total. Trastuzumab: The first cycle dose is 8mg/kg, and each subsequent cycle is 6mg/kg, iv, Day 1, q3weeks, a total of 6 cycles.
  Interventions: Drug: Pyrotinib combined with albumin-bound paclitaxel and trastuzumab

INTERVENTIONS:
Drug: Pyrotinib combined with albumin-bound paclitaxel and trastuzumab — Pyrotinib: 400mg, po,qd,with warm water within 30 minutes after breakfast, q3weeks, 6 cycles in total. Albumin-bound paclitaxel: 260mg/m2, iv, Day1, q3weeks, 6 cycles in total. Trastuzumab: The first cycle dose is 8mg/kg, and each subsequent cycle is 6mg/kg, iv, Day 1, q3weeks, a total of 6 cycles.

SUMMARY:
This study aimed to evaluate the Pyrotinib in combination with albumin-bound paclitaxel and trastuzumab to neoadjuvant therapy efficacy and safety of Her2-positive early or locally advanced breast cancer

DETAILED DESCRIPTION:
Subjects who met the criteria for admission were treated with pyrotinib combined with albumin-bound paclitaxel and trastuzumab (q3w) neoadjuvant therapy for 6 cycles before surgery, and DCR and ORR were assessed before surgery.All subjects who are suitable for surgery undergo surgery and evaluate their pCR rate (pathological complete remission rate).After the operation, the subjects received adjuvant chemotherapy of epirubicin hydrochloride + cyclophosphamide (q3w) for 4 cycles, and at the same time, according to the researcher's recommendation, they chose the follow-up anti-HER2 treatment plan: it is recommended that subjects who have achieved pCR receive preoperative the same anti-Her2 treatment for 1 year; for non-pCR subjects, T-DM1 or trastuzumab and Pertuzumab can be used for anti-her2 treatment for 1 year.For subjects whose estrogen receptor (ER) and/or progesterone receptor (PR) are positive, endocrine therapy can be started at the end of adjuvant chemotherapy.If there are clinical indications at the end of adjuvant chemotherapy, radiotherapy can be given.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18 to 70 who were newly treated.
2. ECOG systemic state 0~1.
3. According to the RECIST 1.1 , at least one measurable lesion exists.
4. Patients with HER2-positive breast cancer confirmed by pathological examination, clinical stage II-III [cT2 and any N, cT3 and any N; cT4 and any N, according to American Joint Committee on Cancer (AJCC) standards] Note: HER2 positive means that the result of the pathology department of the participating center hospital is positive, which is defined as the immunohistochemistry (IHC) test result is 3+ or the in situ hybridization (ISH) result is HER2 gene amplification (HER2/CEP17≥2.0 or Average HER2 copy number/cell ≥6).
5. The functional level of organs must meet the following requirements: 1) Blood routine: ANC≥1.5×109/L; PLT≥90×109/L; Hb≥90 g/L; 2) Blood biochemistry: TBIL≤1.5×ULN; ALT and AST≤2×ULN; BUN and Cr≤1.5×ULN and creatinine clearance ≥50 mL/min (Cockcroft-Gault formula); 3) Heart color Doppler ultrasound: LVEF≥50%; 4) 12-lead ECG: Fridericia corrected QT interval (QTcF) female <470 ms.
6. The hormone receptor status is known.
7. The serum pregnancy test is negative and patients with reproductive potential must agree to use effective non-hormonal contraceptive methods during treatment and at least 6 months after the last use of the test drug.
8. Volunteer to join the study, sign informed consent, have good compliance and are willing to cooperate with follow-up.

Exclusion Criteria:

1. Patients with inflammatory breast cancer.
2. Patients with metastatic breast cancer (stage IV).
3. Inability to swallow, chronic diarrhea and intestinal obstruction, as well as other factors that affect the administration and absorption of the drug.
4. At the same time receive anti-tumor therapy in other clinical trials, including endocrine therapy, bisphosphonate therapy or immunotherapy.
5. Have received major surgery not related to breast cancer within 4 weeks before enrollment, or have not fully recovered from the surgery.
6. Previously used or currently using anti-HER2 targeted drugs (including trastuzumab, pertuzumab, lapatinib, neratinib and pirotinib, etc.).
7. Suffered from other malignant tumors in the past 5 years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma.
8. Accept any other anti-tumor therapy at the same time.
9. Those who are known to have a history of allergies to the drug components of this program; have a history of immunodeficiency, including a positive HIV test, or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation.
10. Previously suffering from heart diseases, including: (1) angina pectoris; (2) arrhythmia requiring medication or clinical significance; (3) myocardial infarction; (4) heart failure; (5) judged by the investigator other heart diseases that are not suitable for participating in this trial.
11. Female patients during pregnancy and lactation;The pregnancy test is positive;Female patients of childbearing age who are unwilling to take effective contraceptive measures during the trial.
12. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study (including but not limited to severe hypertension that cannot be controlled by drugs, severe diabetes, active infection, etc.).
13. Have a clear history of neurological or psychiatric disorders, including epilepsy or dementia.
14. Concomitant use of CYP3A4 inhibitors or inducers.
15. The investigator judges that it is not suitable to participate in any other situations in this research.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) (ypT0/is N0) | Estimated up to 2.5 year
  No microscopically detectable remnants of aggressive tumors in breast and axillary lymph nodes, ductal carcinoma in situ is allowed

SECONDARY OUTCOMES:
Objective response rate (ORR) | Estimated up to 2.5 year
  The percentage of subjects with CR or PR as the best response during the period from the beginning of the treatment to the progression of the disease or the completion of preoperative neoadjuvant therapy 【(CR+PR)/Analysis of the total number of people】.The solid tumor response assessment standard (RECIST 1.1 standard) was used to assess the objective tumor response.
Disease Control Rate (DCR) | Estimated up to 2.5 year
  The percentage of patients with complete remission (CR), partial remission (PR) and stable disease (SD) (≥4 weeks) confirmed by the RECIST 1.1 standard among patients with evaluable efficacy.
Complete remission rate of breast pathology (bpCR） | Estimated up to 2.5 year
  No microscopically detectable remnants of aggressive tumors in breast, ductal carcinoma in situ is allowed
Adverse events (AEs) [ Time Frame: From screening phase until AEs returns to Grade 0-1 or baseline ] | Estimated up to 2.5 year
  AEs were graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
  In general, AEs are graded according to the following: Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE.
  The type, grade and frequency of AEs will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Luo, post-doctor, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Chengdu, Sichuan, China, China

IPD SHARING:
Plan to Share IPD: No